CLINICAL TRIAL: NCT05242705
Title: Serum Cysteine Rich Protein 61 and Cystatin C for Early Detection of Acute Kidney Injury in Patients With Acute Coronary Syndromes
Brief Title: Serum Cysteine Rich Protein 61 and Cystatin C for Early Detection of Acute Kidney Injury in Patients With Heart Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrook S. Ahmed, principal investigator, Assiut University
Other Study IDs: SHSAS
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum Cysteine Rich Protein 61 — collection of serum samples for chemical analysis
  Other Names: Serum Cystatin C

SUMMARY:
Acute Kidney Injury (AKI) is defined as an absolute increase in serum creatinine ≥0.3 mg/dl (≥26.4 μmol/l), a percentage increase in serum creatinine ≥50% (1.5-fold from baseline), or a reduction in urine output (documented oliguria < 0.5 ml/kg/hour for > 6 hours) S.creatinine which is considered the gold standard currently for diagnosis of AKI remains unchanged until 50% of kidney function falls down. It is affected by non-specific factors like diet, age, dehydration, muscle mass, gender, and drugs.

There were evidences of the association between AKI and acute coronary syndrome (ACS); First, AKI detection may be missed by cardiologists. Physicians tend to disregard mild or transient serum creatinine elevation during hospital stay for ACS, and they often attribute small serum creatinine increases to laboratory variations.

DETAILED DESCRIPTION:
Cystatin C (CysC), a cystatin protease inhibitor, is less affected by non-specific factors. When glomerular filtration rate (GFR) decreases, CysC begins to increase.

CysC was recommended to be measured in addition to creatinine in GFR estimation.

Cysteine-rich protein 61 (Cyr61) is a cysteine-rich secretory protein that promotes cell proliferation, adhesion, chemotaxis, embryonic development and neovascularization . Previous studies have detected low expression level of Cyr61 in normal adult kidney and high expression of Cyr61 in ischemic rats and mice kidney, which suggests that Cyr61 may be a potential biomarker for diagnosis of AKI . CYR61 might possibly identify patients with more severe kidney injury, which would be very beneficial for early treatment of AKI after

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Informed consent
3. Patient with absolute increase in serum creatinine ≥0.3 mg/dl (≥26.4 μmol/l) or with percentage increase in serum creatinine ≥50% (1.5-fold from baseline)
4. Patient with reduction in urine output (documented oliguria < 0.5 ml/kg/hour for > 6 hours)
5. Patient with typical chest pain, ECG changes, Echocardiogram positive finding

Exclusion Criteria:

1. History of nephrectomy
2. patient with renal transplantation
3. patient with renal replacement therapy initiated before admission
4. patient with chronic kidney disease
5. patient on regular haemodialysis
6. patient known to be diabetic

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient come to assuit university hospital with typical chest pain, ECG changes, Echocardiogram positive finding then develope absolute increase in serum creatinine ≥0.3 mg/dl (≥26.4 μmol/l), with percentage increase in serum creatinine ≥50% (1.5-fold from baseline) or with reduction in urine output (documented oliguria < 0.5 ml/kg/hour for > 6 hours)
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Early detection of acute kidney injury in patient with acute coronary syndromes after cardiac interventional surgeries as primary percutaneous coronary intervention (PCI) | 3 years
  Early detection of acute kidney injury in patient with acute coronary syndromes after cardiac interventional surgeries as primary percutaneous coronary intervention (PCI)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marenzi G, Cosentino N, Bartorelli AL. Acute kidney injury in patients with acute coronary syndromes. Heart. 2015 Nov;101(22):1778-85. doi: 10.1136/heartjnl-2015-307773. Epub 2015 Aug 4. PMID 26243789
- [Background] Zhang Z, Lu B, Sheng X, Jin N. Cystatin C in prediction of acute kidney injury: a systemic review and meta-analysis. Am J Kidney Dis. 2011 Sep;58(3):356-65. doi: 10.1053/j.ajkd.2011.02.389. Epub 2011 May 20. PMID 21601330
- [Background] Shlipak MG, Mattes MD, Peralta CA. Update on cystatin C: incorporation into clinical practice. Am J Kidney Dis. 2013 Sep;62(3):595-603. doi: 10.1053/j.ajkd.2013.03.027. Epub 2013 May 20. PMID 23701892
- [Background] Mosa OF, Skitek M, Kalisnik JM, Jerin A. Evaluation of serum cysteine-rich protein 61 and cystatin C levels for assessment of acute kidney injury after cardiac surgery. Ren Fail. 2016 Jun;38(5):699-705. doi: 10.3109/0886022X.2016.1157747. Epub 2016 Mar 16. PMID 26982887